CLINICAL TRIAL: NCT06919718
Title: Effects of Maternal Stress on Human Milk Composition and Subsequent Infant Outcomes
Brief Title: Impact of Vitamin D Supplements on Mental Health and Milk Composition in Mothers Living in Idaho
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB 20-024; P20GM152304 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Maternal Stress
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Control (Placebo Comparator)
  Interventions: Other: Placebo
- Vitamin D (Experimental)
  Interventions: Dietary Supplement: Vitamin D (Cholecalciferol )

INTERVENTIONS:
Dietary Supplement: Vitamin D (Cholecalciferol ) — 2,000 IU Vitamin D
  Arms: Vitamin D
Other: Placebo — Placebo
  Arms: Placebo Control

SUMMARY:
Mothers of preterm infants experience exaggerated emotional stressors compared to those typically associated with new motherhood, making these women particularly vulnerable to postpartum depression. As many as 70% of mothers of preterm infants experience postpartum depression compared to only 12.5% of those delivering full-term infants. Increased stress and depression during this critical period are detrimental because they hamper a mother's ability to care for her infant and are associated with increased neonatal sepsis and mortality, decreased neonatal growth, and delayed motor and cognitive development. Postpartum depression is also associated with excessive maternal weight gain and risk for metabolic diseases, anxiety, and sleep disturbances. Stress in breastfeeding mothers can also alter circulating concentrations of some bioactive components (e.g., immunoglobulins, cortisol) that can transfer into milk. As such, understanding factors predisposing these vulnerable women to extreme levels of stress and finding ways to lower this stress and lessen its negative health outcomes on mothers and infants are important public health challenges. The March of Dimes estimates that 8.5% of births in Idaho are preterm, making this topic particularly relevant for Idaho women. Risk factors for postpartum depression in mothers delivering term or preterm infants are complex, but maternal nutrient deficiencies may be involved. Vitamin D status, for instance, is inversely correlated with risk of postpartum depression in women delivering term infants. However, vitamin D interventions have yielded inconsistent results, perhaps due to confounding impacts of geographic location, skin color, and endogenous vitamin D synthesis. Endogenous vitamin D synthesis requires cutaneous sunlight exposure, placing Idaho women at even greater risk of vitamin D deficiency - particularly in the winter when days are extremely short (only 7 hr on the winter solstice). The impact of maternal vitamin D supplementation during lactation on infant variables (e.g., vitamin D status) has been examined. However, its effect on maternal mental health has not been rigorously studied - let alone in the 'frontier and remote' (FAR) rural West, including Idaho, with short periods of wintertime sunlight and poor access to healthcare. Our long term goal is to develop interventions to improve maternal and infant health in Idaho - particularly in the context of preterm births. The overall primary objective of this proposal is to determine if maternal vitamin D supplementation improves vitamin D status and mental health in Idahoan mothers of preterm infants. Our central hypothesis is that vitamin D supplementation improves vitamin D status and reduces stress and other indicators of poor postpartum maternal mental health in Idaho women delivering preterm infants. Secondarily, we will assess the effects of maternal vitamin D supplementation on human milk composition.

ELIGIBILITY:
Inclusion Criteria:

* Mothers (>/= 18 years of age) of newborn infants (within first 4 months postpartum) in Idaho

Exclusion Criteria:

* Mothers (<18 years of age) of newborn infants (within first 4 months postpartum)
* Infants not anticipated to survive >72 hours

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Stress | baseline, 4-week, 8-week
  Maternal stress measured by the validated questionnaire: Perceived Stress Scale (PSS).
  The PSS can range from 0 to 40 with higher scores indicating higher perceived stress:
  0-13 = low stress 14-26 = moderate stress 27-40 = high stress
Maternal Depression | baseline, 4-week, 8-week
  Maternal depression measured using the validated questionnaire: Edinburgh Postnatal Depression Scale.
  The Edinburgh Postnatal Depression Scale can range from 0 to 30 with higher scores indicating higher depression. Any total score >10 indicates depression.
Maternal Vitamin D status | baseline, 4-week, 8-week
  Blood vitamin D concentration

SECONDARY OUTCOMES:
Maternal Self-Compassion | 8-week
  Maternal self-compassion measured using the validated Self-Compassion-Short Form
Maternal physiologic stress | baseline, 4-week, 8-week
  Blood and salivary cortisol
Physiologic Maternal Self-compassion | baseline, 4-week, 8-week
  Blood oxytocin concentrations
Milk Immunomodulatory Composition | baseline, 4-week, 8-week
  Milk Immunomodulatory protein concentrations

OTHER OUTCOMES:
Maternal Diet | baseline, 4-week, 8-week
  Diet assessed using 24-hour diet recall

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kootenai Health, Coeur d'Alene, Idaho
  - University of Idaho, Moscow, Idaho